CLINICAL TRIAL: NCT02567786
Title: Comparison of Fresh Frozen Plasma and Plasmalyte ® for Priming Cardiopulmonary Bypass in Infants and Children Undergoing Open-heart Surgery: A Double-blind Randomized Controlled Study
Brief Title: Fresh Frozen Plasma and Plasmalyte ® for Priming Cardiopulmonary Bypass in Infants and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Mona Momeni, MD, PhD, Clinical Professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Plasma versus Plasmalyte
Record Dates: First submitted 2015-09-29; First posted 2015-10-05 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Surgical Procedures, Operative; Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Fresh Frozen Plasma (Active Comparator): The priming of the CPB oxygenator will be done with 15 ml/kg of FFP in addition to packed red blood cells.
  Interventions: Procedure: Surgery with CPB; Other: Fresh Frozen Plasma
- Plasmalyte (Active Comparator): The priming of the CPB oxygenator will be done with 15 ml/kg of Plasmalyte in addition to packed red blood cells.
  Interventions: Procedure: Surgery with CPB; Other: Plasmalyte

INTERVENTIONS:
Procedure: Surgery with CPB
Other: Fresh Frozen Plasma
  Arms: Fresh Frozen Plasma
Other: Plasmalyte
  Arms: Plasmalyte

SUMMARY:
Coagulation abnormalities after pediatric open-heart surgery are complex and very often multifactorial. Besides the cardiopulmonary bypass (CPB), the congenital pathology and the coagulation tests during CPB, the younger age has been the most significant risk factor for bleeding and transfusion requirements. In children the volume of pump priming is much higher compared with the patient's circulating blood volume. For this reason the CPB tubing system is primed with packed red blood cells and fresh frozen plasma (FFP) to avoid excessive hemodilution and induced coagulopathy. While this is routinely performed in neonates and small infants, the routine priming of CPB system with FFP has been questioned in several randomized prospective studies in older infants. However, the results of these studies are conflicting. Moreover, they show methodological issues.

ELIGIBILITY:
Inclusion Criteria:

* Children weighing between 7 and 15 kg and admitted to undergo open-heart surgery with CPB

Exclusion Criteria:

* Patients with preoperative coagulation abnormalities
* Parental refusal
* Emergency surgery
* Patients with preoperative renal or hepatic dysfunction

Ages: 2 Months to 70 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Postoperative bleeding (mL blood in the chest tubes). Significant postoperative bleeding is defined as a bleeding of > 5ml/kg/h in the first 6hours postoperatively. | The first 6 hours postoperatively
  The exact amount of blood loss in the postoperative period per kilogram weight of child.
Increased risk of of donor exposure intraoperatively and postoperatively. | The first 6 hours postoperatively
  The total number of different packs of allogeneic blood products administered per child.

SECONDARY OUTCOMES:
Volume of transfused allogenic blood products (mL). | The first 6 hours postoperatively
  The total volume of allogeneic blood products per kilogram weight of child.
Comparison of Rotem and Multiplate between both groups. | The first 6 hours postoperatively
  The results of the point-of-care tests ROTEM and Multiplate will be compared between children in the Plasmalyte group and children in the Fresh Frozen Plasma group.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Momeni, MD,PhD, Principal Investigator — Université Catholique de Louvain; Cliniques Universitaires Saint Luc
Locations (1):
- Mona Momeni, Brussels, Belgium